CLINICAL TRIAL: NCT02521532
Title: Dietary Nitrate for COPD: a 14d, Randomized, Placebo-controlled, Crossover Trial
Brief Title: A 2 Week, Crossover Trial of Dietary Nitrate in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: University College Dublin (Other); Connolly Hospital Blanchardstown (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Chronic NO3- in COPD
Record Dates: First submitted 2015-01-07; First posted 2015-08-13 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitrate rich beetroot juice (Experimental): Concentrated, beetroot juice is a rich source of dietary nitrate.
  Interventions: Dietary Supplement: Dietary nitrate
- Nitrate depleted placebo beetroot juice (Placebo Comparator): Placebo beetroot juice is identical to active beetroot juice in every way except nitrate content.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Dietary nitrate — 140ml of nitrate rich beetroot juice provides 12.9mmol nitrate and will be consumed on a daily basis during the intervention by the study subjects.
  Other Names: Beetroot juice
  Arms: Nitrate rich beetroot juice
Dietary Supplement: Placebo — 140ml of nitrate depleted beetroot juice provides 0.5mmol nitrate and will be consumed on a daily basis during the intervention by the study subjects.
  Other Names: Nitrate depleted beetroot juice
  Arms: Nitrate depleted placebo beetroot juice

SUMMARY:
Acute consumption of dietary nitrate (as beetroot juice) has been shown to increase exercise and decrease systemic blood pressure in multiple populations, including COPD. The chronic effect of dietary nitrate in obstructive sleep apnea syndrome (OSAS) has not been reported.

DETAILED DESCRIPTION:
Acute consumption of dietary nitrate (as beetroot juice) has been shown to increase exercise and decrease systemic blood pressure in multiple populations, including COPD. The chronic effect of dietary nitrate in OSAS has not been reported.

The investigators hypothesize that chronic nitrate consumption might increase exercise tolerance, and exhaled NO but decrease blood pressure and have little impact on quality of life and pulmonary function.

This study is a randomized, double-blind placebo-controlled, crossover trial. At baseline, mid-point and endpoint exercise tolerance, pulmonary function, quality of life and ambulatory blood pressure will be assessed in conjunction with demographics and blood draw. After baseline measures, each subject will be randomized to consume nitrate rich beetroot juice for 14 consecutive nights when assessments will be repeated followed by 14 nights of placebo and endpoint assessments or the converse.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable,
* Diagnosed with COPD
* Ambulatory out-patients

Exclusion Criteria:

* Long term oxygen therapy
* Pulmonary hypertension
* Active cardiovascular disease
* Active skeletal conditions
* Taking vasodilators
* Diabetes mellitus

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in incremental shuttle walk test distance | Day 1, day 15 and day 29

SECONDARY OUTCOMES:
Change in plasma nitrate | Day 1, day 15 and day 29
  Assessed by chemiluminescence
Change in ambulatory blood pressure | Day 1, day 15 and day 29
Change in quality of life | Day 1, day 15 and day 29
  Quality of Life will be assessed with the Clinical COPD Questionnaire
Change in forced expiratory volume | Day 1, day 15 and day 29
  Assessed by spirometry
Change in inflammatory markers | Day 1, day 15 and day 29
  Assessed by C-reactive protein
Change in forced vital capacity | Day 1, day 15 and day 29
  Assessed by spirometry
Change in plasma nitrate and nitrite | Day 1, day 15 and day 29
  Assessed by chemiluminescence

CONTACTS AND LOCATIONS:
Overall Officials: Liam Cormican, MD, Principal Investigator — Respiratory & Sleep Diagnostics Department, Connolly Hospital, Dublin 15, Ireland
Locations (1):
- Respiratory & Sleep Diagnostics Department, Connolly Hospital, Dublin, Ireland